CLINICAL TRIAL: NCT02618954
Title: Value of Ultrasound for Evaluating Rheumatoid Arthritis in Remission: Longitudinal Study
Brief Title: Role of Ultrasound for Evaluating Rheumatoid Arthritis in Remission
Acronym: SONORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9186
Record Dates: First submitted 2015-11-19; First posted 2015-12-02 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Rheumatoid Arthritis in Remission
Keywords: Rheumatoid arthritis; Articular ultrasound; Synovitis; Relapse risk
MeSH Terms: conditions — Arthritis, Rheumatoid; Synovitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study patient (Other): Articular ultrasound at each study follow-up
  Interventions: Other: Articular ultrasound

INTERVENTIONS:
Other: Articular ultrasound — (Device : Ultrasound) : Articular ultrasound of the Disease Activity Score (DAS) 28 articular joint

SUMMARY:
The objective of this study is to determine the longitudinal relation between clinical remission and ultrasound (US) remission in Rheumatoid arthritis (RA).

At a patient level, US-detected residual synovitis (evaluated both by US grey-scale signals and power Doppler signals) is frequent in patients with RA in clinical remission. Several longitudinal studies reveal an association of US-detected residual synovitis and risk of relapse and radiographic progression, in individual patients and joints, over 1-2 years.

However, the longitudinal relation between clinical remission and US remission is not so well-known and it is possible that clinical remission arrive before ultrasound remission. Thus arise the question as to whether the presence of US-detected residual synovitis require to adapt the treatment to ultrasound findings or to simply increase the patient care.

The investigator propose to conduct a prospective, bi-center, non randomized study.

DETAILED DESCRIPTION:
The study population will include all RA patient at least 18 years old in clinical remission for less than 6 month.

The primary endpoint (ability of US-detected residual synovitis to predict relapse or radiographic progression in individual patients and joints) will be evaluated afer 12 months of follow-up The total follow-up will be 12 months with a follow-up every 3 months. In addition to the standard care, each follow-up will include an ultrasound examination of 40 joints and 8 tendons

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* PR fulfilling ARC / EULAR (European League Against Rheumatism) 2010 criteria
* Patient treated by DMARDs (disease-modifying antirheumatic drug)
* Patient in confirmed remission for less than 6 months

Exclusion Criteria:

* Patient participating simultaneously in another clinical study with blind treatment
* Patient participating simultaneously in another clinical study involving decreasing of drug dose
* Patient in post clinical study exclusion period
* patients subject to legal protection measures
* Patient unable to read French
* Pregnant or breast-feeding women
* patient treated with Rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
1 year pejorative evolution | 1 year after inclusion
  Number of patient with a clinical relapse

SECONDARY OUTCOMES:
Structural progression | 1 year after inclusion
  Number of patient with a structural progression of the illness
RA (Rheumatoid Arthritis) remission duration | At each follow-up (3,6,9 and 12 months after inclusion)
  Evaluation of the remission duration (patient in both clinical and ultrasound remission)
RA ultrasound remission duration | At each follow-up (3,6,9 and 12 months after inclusion)
  Evaluation of the ultrasound remission duration
RA clinical remission duration | At each follow-up (3,6,9 and 12 months after inclusion)
  Evaluation of the clinical remission duration
Clinical relapse at one year | 1 year after inclusion
  Evaluation of the probability of a clinical relapse at 1 year based on the ultrasound data
Persistence of ultrasound synovitis (lenght of RA evolution, lenght of clinical remission, anti-CCP, biological inflammatory symptom persistence, treatments) | At baseline
  identifying initial factors that can explain persistence of ultrasound synovitis despite clinical remission
Radiographic progression at 1 year | 1 year after inclusion
  Evaluation at joint level the probability of a radiographic progression in presence of a non active synovitis
Intra-observator reproductibility | 1 year after inclusion
  Evaluating the intra-observer reliability for US synovitis through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Gaël Mouterde, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, Herault, France